CLINICAL TRIAL: NCT01493856
Title: A Randomized, Open Label, Single-Dose, 2-Way Cross-over Clinical Trial to Compare the Safety and Pharmacokinetic Characteristics of Combination of Rosuvastatin and CS-866 and DWJ1276 in Healthy Male Volunteers
Brief Title: A Clinical Trial to Compare the Safety and Pharmacokinetic Characteristics of Combination of Rosuvastatin and CS-866 and DWJ1276
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DW_DWJ1276002
Record Dates: First submitted 2011-12-13; First posted 2011-12-16 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Olmesartan Medoxomil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin+Olmesartan (Active Comparator): single dose of Rosuvastatin 20mg and olmesartan medoxomil(CS-866) 40mg
  Interventions: Drug: Cresto; Drug: Olmetec
- DWJ1276 (Experimental): Single dose of DWJ1276
  Interventions: Drug: DWJ1276

INTERVENTIONS:
Drug: Cresto — tablet, rosuvastatin 20mg
  Arms: Rosuvastatin+Olmesartan
Drug: Olmetec — tablet, olmesartan medoxomil(CS-866) 40mg
  Arms: Rosuvastatin+Olmesartan
Drug: DWJ1276 — tablet, Rosuvastatin 20mg and olmesartan medoxomil 40mg
  Arms: DWJ1276

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetic characteristics of combination of rosuvastatin and CS-866 and DWJ1276 alone.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male volunteers aged 20 to 50 years
2. A subject who provided written informed consent to participate in this study and cooperative with regard to compliance with study related constraints

Exclusion Criteria:

1. A subject who had any allergic history to any drug.
2. A subject with sign or symptoms or previously diagnosed disease of liver, kidney, neurology, respiratory, endocrinology, hematology, cardiovascular, genitourinary, psychology, ophthalmic, dermatology and gastrointestinal function or other significant diseases
3. History or suspicion of current drug abuse
4. A subject who had received treatment with below listed drug within specified period prior to the first dose of study medication

   * Within 1 month: drug known CYP inducer or inhibitor
   * Within 2 weeks: Prescribed or herbal medicine
   * Within 1 weeks: OTC medicine
   * Within 2 days: Consumption of caffeine
5. A subject who had participated in any other clinical study within the last 2 weeks
6. A subject from whom over 400mL of blood was sampled(whole blood donation) within last 2 weeks or plasma/platelet donation within 1 month.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
AUClast | 18 time points up to 72 hours
Cmax | 18 time points up to 72 hours

SECONDARY OUTCOMES:
AUCinf | 18 time points up to 72 hours
T1/2 | 18 time points up to 72 hours
%AUCextra | 18 time points up to 72 hours
Tmax | 18 time points up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kyungsoo Park, M.D., Ph.D., Principal Investigator — YONSEI UNIVERSITY HEALTH SYSTEM (YUHS)
Locations (1):
- Yonsei University Health System (Yuhs), Seoul, South Korea